CLINICAL TRIAL: NCT03256630
Title: A Laboratory Study To Evaluate A Blood Biomarker That Can Distinguish Between the Presence Or Absence of Aggressive Prostate Cancer
Brief Title: Evaluation of a Blood Biomarker to Try and Distinguish Between the Presence or Absence of Aggressive Prostate Cancer
Status: Terminated | Type: Observational
Why Stopped: Business decision to discontinue development of the IsoPSA assay.
Sponsor: Genomic Health®, Inc. (Industry)
Collaborators: AdventHealth (Other)
Responsible Party: Sponsor
Other Study IDs: 09-048
Record Dates: First submitted 2017-08-16; First posted 2017-08-22 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Prostate Cancer
Keywords: Active Surveillance; Radical Prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Blood, Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A Laboratory Study to Evaluate Urine and Blood Biomarkers That Can Distinguish Between the Presence or Absence of Aggressive Prostate Cancer

DETAILED DESCRIPTION:
The over-arching goal of this study is to evaluate if biomarkers within the blood or urine of men with localized prostate cancer can distinguish between those with indolent cancer, defined as Gleason Grade Groups 1 and 2 and those with more aggressive disease (Gleason Grade Groups 3, 4, and 5).

ELIGIBILITY:
Inclusion Criteria:

1. Patient has been diagnosed with Prostate Cancer and is planning on having a Radical Prostatectomy performed at the Global Robotics Institute.
2. Diagnostic PSA ≤ 20 ng/mL.
3. Pathology report from most recent positive biopsy, prior to Radical Prostatectomy, is available.
4. Ability to read and understand the informed consent form.
5. Patient must have signed informed consent form

Exclusion Criteria:

1. Any of the following active therapies received: radiation, chemotherapy, biologic agents, surgery, local therapies including cryotherapy or HIFU.
2. Diagnostic PSA > 20 ng/mL or missing PSA.
3. Patients who are unable or unwilling to provide informed consent.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Prostate cancer patients who are planning to have a Radical Prostatectomy at the Global Robotics Institute and are informed and willing to participate in study.
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Characterize the distribution of clinical/pathological factors of the samples by the Gleason Grade Group and to characterize the distribution of the signal of each biomarker by the Gleason Grade Group or combination of groups. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Florida Hospital Global Robotics Institute, Celebration, Florida, United States